CLINICAL TRIAL: NCT04458402
Title: Phase I Study of Adjuvant Hypofractionated Whole Pelvis Radiation Therapy in Endometrial Cancer.
Brief Title: Adjuvant Hypofractionated Whole Pelvis Radiation Therapy in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teresa Meier (Other)
Responsible Party: Sponsor-Investigator, Teresa Meier, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-GYN-20-01
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose allocation will be based upon a Bayesian continual reassessment method that incorporates patient-reported outcomes (PRO-CRM17), which uses separate models for the probability of C-DLT and the probability of P-DLT, as well as the accumulated C-DLT and P-DLT data at each dose level, to sequentially allocate each new patient cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hypofractionated Whole-Pelvis Radiotherapy (Experimental): Hypofractionated WPRT Cohort 1: 41.25 Gy in 15 fx Cohort 2: 38 Gy in 10 fx
  Interventions: Radiation: Hypofractionated WPRT

INTERVENTIONS:
Radiation: Hypofractionated WPRT — Cohort 1: 41.25 Gy in 15 fx Cohort 1: 38 Gy in 10 fx

SUMMARY:
Studying adjuvant hypofractionated whole pelvis radiation therapy in Endometrial Cancer.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety of adjuvant hypofractionated whole pelvis radiation therapy (WPRT) in endometrial cancer. The primary objective of the study is to determine the maximum tolerated dose per fraction (MTDF), defined by acceptable acute clinician-reported GI and GU toxicity and patient-reported GI toxicity, of WPRT from among the two study dose levels. Acute GI and GU toxicity will be assessed according to both the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0, and Patient Reported Outcome-CTCAE (PRO-CTCAE). Clinician-reported dose-limiting toxicity (C-DLT) is a binary outcome (yes/no), defined as an acute grade 3 or higher GI or GU per CTCAE, occurring within three months of completing WPRT. Patient-reported DLT (P-DLT) is a binary outcome, defined by a GI toxicity with a score of ≥4 on the 5-point scale per PRO-CTCAE, occurring within three months of completing WPRT. The MTDF is defined as the minimum of the dose with a C-DLT rate closest to the clinician-reported target C-DLT rate of 20% and the dose with a P-DLT rate closest to the patient-reported target P-DLT rate of 55%. Toxicity results of NRG-RTOG 1203- A Randomized Phase III Study of Standard vs. IMRT Pelvic Radiation for Post-Operative Treatment of Endometrial and Cervical Cancer- were used to define the acceptable percentage of DLTs. The study will accrue participants in cohorts of size 3. The starting dose level will be dose level 1 (41.25 Gy in 15 fx).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed stage I, II, or III endometrial cancer who require pelvic radiation as determined by their treating radiation oncologist and/or gynecologic oncologist. Patients may also be identified through the Gynecologic Oncology Multidisciplinary Tumor Board. The decision to include Stage I patients will be based on risk factors for recurrence including tumor grade, extent of myometrial invasion, presence of lymphovascular space invasion, and histology (endometrioid, papillary serous, clear cell, carcinosarcoma). Stage I patients may include those who are ineligible for vaginal cuff brachytherapy due to patient anatomy or those who are at higher risk for pelvic nodal recurrence and pelvic external beam radiotherapy is preferred over vaginal cuff brachytherapy.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Patients must have undergone total hysterectomy and bilateral salpingo-oophorectomy with or without pelvic and/or para-aortic lymph node dissection/sampling or sentinel lymph node (SLN) dissection.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with an Inflammatory Bowel Disease diagnosis, regardless of disease activity.
* Patients with current, active disease involving periaortic node(s). This is based on histologically positive para-aortic node(s) removed at time of surgery.
* Patients with gross residual disease following surgical resection. Final pathologic margins must be negative (no tumor on ink). This may also be determined clinically by the gynecologic oncologist at time of surgery or post-operative imaging if applicable. Post-operative imaging is not required at time of surgery.
* Patients who have ever had pelvic radiotherapy prior to entering the study.
* Patients who are receiving any other investigational agents. Patients who have received other investigational agents previously who are no longer receiving these investigational agents may be eligible at the discretion of the PI.
* Patients with uncontrolled intercurrent illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 8 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Safety profile of hypofractionated, isoeffective whole pelvis radiation regimens for post-operative treatment of endometrial cancer using CTCAE version 5.0 and Patient Reported Outcome-CTCAE. | 3 months
  Toxicity profile will be determined by assessment of acute gastrointestinal and genitourinary toxicity during WPRT and 3 months post-radiation using CTCAE version 5.0 and Patient Reported Outcome-CTCAE (PRO-CTCAE). Dose-limiting toxicity (DLT) will be defined as any acute ≥ grade 3 gastrointestinal or genitourinary per CTCAE or a score of ≥4 on the 5-point scale per PRO-CTCAE.
Maximum tolerated dose per fraction (MTDF) of hypofractionated, isoeffective whole pelvis radiation regimens for post-operative treatment of endometrial cancer through CTCAE data and gastrointestinal PRO-CTCAE data. | 3 months
  Determination of the MTDF will rely on toxicity data, specifically combined gastrointestinal and genitourinary CTCAE data and gastrointestinal PRO-CTCAE data. MTDF should not exceed >20% of patients having a DLT per CTCAE or >55% of patients having a dose-limiting GI toxicity per PRO-CTCAE. Further details in study design.

SECONDARY OUTCOMES:
Impact of hypofractionated WPRT on patient quality of life using the Functional Assessment of Cancer Therapy-Endometrial version 4.0. | 3 months
  Quality of life data will be obtained for exploratory analysis only.
Patient compliance with hypofractionated WPRT, as defined by how many patients are able to complete WPRT without a break in treatment. | 3 months
  Patient compliance with radiotherapy will be recorded and used for exploratory analysis only.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Meier, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wages NA, Nelson B, Kharofa J, Meier T. Application of the patient-reported outcomes continual reassessment method to a phase I study of radiotherapy in endometrial cancer. Int J Biostat. 2022 Nov 17;19(1):163-176. doi: 10.1515/ijb-2022-0023. eCollection 2023 May 1. PMID 36394530